CLINICAL TRIAL: NCT03666897
Title: Markers of Recovery in StrokE Study
Brief Title: Markers of Recovery in StrokE Study (MORSE)
Acronym: MORSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-016
Record Dates: First submitted 2018-08-07; First posted 2018-09-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTI Outcomes and Biomarkers (Other): Imaging and Lab Collection
  Interventions: Other: DTI Images and Plasma Biomarkers

INTERVENTIONS:
Other: DTI Images and Plasma Biomarkers — Additional Images added from standard of care MRI, Bio-markers identified

SUMMARY:
Our current biological understanding of stroke recovery in humans is extremely limited and this lack of knowledge is a major challenge in reducing stroke disabilities and deficits. Evidence of neural repair in humans can be gleaned indirectly through functional outcome measures, but we propose that metabolomics may also provide a minimally invasive window into human brain repair. This study will integrate clinical imaging and molecular biomarkers as a diagnostic tool in further understanding stroke recovery mechanisms.

DETAILED DESCRIPTION:
Our long-term goal is to improve and hasten recovery following a stroke with translational research, which would combine the use of neuroimaging and identify neural repair metabolites. The objective and sequential step in fulfilling our long-term goal, is to identify differential expression of select stroke plasma biomarkers of neural repair, and image CST integrity in patients with good and poor recovery following an ischemic stroke. Diffusion tension imaging (DTI), will be used to image the neural repair as it occurs, further enhancing our understanding of stroke recovery. There are currently no known plasma biomarkers of neural repair. Identification of such biomarkers would be extremely valuable for designing stroke recovery drugs and timing rehabilitation therapies.

ELIGIBILITY:
Inclusion Criteria:

* Imaging confirmed ischemic stroke within 7 days of stroke onset
* Age > 18 years
* NIHSS ≥ 1 on arm item OR NIHSS = 0 on arm item but < 3/5 strength on MRC scale in distal joint (flex/ext elbow or grip/ext hand)
* Pre-stroke modified Rankin Scale (mRS) < 3

Exclusion Criteria:

* Active malignancy (not thought to be cured or in remission)
* Anemia (HCT < 25)
* Sepsis
* Suspected bacterial endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Establish plasma metabolite biomarkers that mirror neuronal repair and identify structural changes following ischemic strokes | 2 years
  Identify differential expression of select stroke plasma biomarkers of neural repair through metabolic testing and imaging CST integrity in patients with good and poor recovery following an ischemic stroke

SECONDARY OUTCOMES:
Change in Fugl-Meyer | Baseline, 90 days post stroke
  The Fugl-Meyer will be used to assess motor function at the shoulder, elbow, wrist, fingers, hip, knee, and foot. The scale ranges from 0 to 66 points, measuring the impairment level of the upper extremity. Zero indicates a high level of impairment or minimum hand motor function, while 66 points indicates an increased motor function which is similar to normal upper extremity function.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Miller, MD, Principal Investigator — Spectrum Health Hospital
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No